CLINICAL TRIAL: NCT00844597
Title: Clinical Study to Assess the Safety fo AVI-4658 in Subjects With Duchenne Muscular Dystrophy Due to a Frame-shift Mutation Amenable to Correction by Skipping Exon 51.
Brief Title: Dose-Ranging Study of AVI-4658 to Induce Dystrophin Expression in Selected Duchenne Muscular Dystrophy (DMD) Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Collaborators: British Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVI-4658-28
Record Dates: First submitted 2008-12-24; First posted 2009-02-16 (Estimated); Results first posted 2015-10-06 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-09

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — eteplirsen; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort 1 - 0.5 mg/kg/wk (Experimental): Subjects in this group will receive a 0.5 mg/kg/wk dose of AVI-4658 over 12 weekly IV infusions in 50 mL of normal saline solution over a 60-minute period
  Interventions: Drug: AVI-4658 for Injection
- Cohort 2 - 1.0 mg/kg/wk (Experimental): Subjects in this group will receive a 1.0 mg/kg/wk dose of AVI-4658 over 12 weekly IV infusions in 50 mL of normal saline solution over a 60-minute period
  Interventions: Drug: AVI-4658 for Injection
- Cohort 3 - 2.0 mg/kg/wk (Experimental): Subjects in this group will receive a 2.0 mg/kg/wk dose of AVI-4658 over 12 weekly IV infusions in 50 mL of normal saline solution over a 60-minute period
  Interventions: Drug: AVI-4658 for Injection
- Cohort 4 - 4.0 mg/kg/wk (Experimental): Subjects in this group will receive a 4.0 mg/kg/wk dose of AVI-4658 over 12 weekly IV infusions in 50 mL of normal saline solution over a 60-minute period
  Interventions: Drug: AVI-4658 for Injection
- Cohort 5 - 10.0 mg/kg/wk (Experimental): Subjects in this group will receive a 10.0 mg/kg/wk dose of AVI-4658 over 12 weekly IV infusions in 50 mL of normal saline solution over a 60-minute period
  Interventions: Drug: AVI-4658 for Injection
- Cohort 6 - 20.0 mg/kg/wk (Experimental): Subjects in this group will receive a 20.0 mg/kg/wk dose of AVI-4658 over 12 weekly IV infusions in 50 mL of normal saline solution over a 60-minute period
  Interventions: Drug: AVI-4658 for Injection

INTERVENTIONS:
Drug: AVI-4658 for Injection — AVI-4658 for Injection, is packaged as 100 mg/mL in phosphate buffered saline with 1 mL per vial. Study dosages will be infused over a 1 hour period with Normal saline in 6 dose cohorts.
  Other Names: Eteplirsen

SUMMARY:
The specific aim of this Phase I/II study is to assess the safety of intravenous administered Morpholino oligomer directed against exon 51 (AVI-4658 PMO).

DETAILED DESCRIPTION:
Primary outcome is safety, tolerability and dose selection for future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed assent (as required by EC) and parents/guardians have provided written informed consent.
2. Has an out-of-frame deletion(s) that could be corrected by skipping exon 51 based on DNA sequencing data from the candidate.
3. Is male and between the ages of ≥ 5 years and ≤ 15 years.
4. Has a muscle biopsy analysis showing < 5% revertant fibres present at baseline.
5. DNA sequencing of the candidate's dystrophin exon 51 confirms that no DNA polymorphisms are present that could compromise PMO duplex formation or there is confirmation of in vitro dystrophin production after AVI-4658 exposure to fibroblast or myoblast in vitro cultures.
6. Intact right and left bicep muscles or alternative arm muscle group.
7. Is able to walk independently at least 25 meters.
8. Has a forced vital capacity (FVC) ≥ 50% of predicted and does not require ventilatory support or supplemental oxygen.
9. Receives the standard of care for DMD as recommended by the DMD care recommendations from the North Star UK and TREAT-NMD.
10. The parent(s) or legal guardian and Subject have undergone counselling about the expectations of this protocol and agree to participate.
11. The parent(s) or legal guardian and Subject intend to comply with all study evaluations and return for all study activities.

Exclusion Criteria:

1. A DNA polymorphism within exon 51 that may compromise PMO duplex formation.
2. Known antibodies to dystrophin.
3. Lacks intact right and left bicep muscles or alternative arm muscle group.
4. A calculated creatinine clearance less than 70% of predicted normal for age based on the Cockcroft and Gault Formula.
5. A left ventricular ejection fraction (EF) of < 35% and/or fractional shortening of <25% based on echocardiography (ECHO)during screening.
6. A history of respiratory insufficiency as defined by need for intermittent or continuous supplemental oxygen.
7. A severe cognitive dysfunction rendering the potential subject unable to understand and comply with the study protocol.
8. Any known immune deficiency or autoimmune disease.
9. A known bleeding disorder or has received chronic anticoagulant treatment within three months of study entry.
10. Receipt of pharmacologic treatment, apart from corticosteroids, that might affect muscle strength or function within 8 weeks of study entry (viz., growth hormone, anabolic steroids).
11. Surgery within 3 months of study entry or planned for anytime during the duration of the study.
12. Another clinically significant illness at time of study entry.
13. Subject or parent has active psychiatric disorder, has adverse psychosocial circumstances,recent significant emotional loss, and/or history of depressive or anxiety disorder that might interfere with protocol compliance.
14. Use of any experimental treatments, has participated in any DMD interventional clinical trial within 4 weeks of study entry or participated in the AVI-4658-33 intramuscular (i.m.) trial.

Ages: 5 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Austen Eddy, MSM, Study Director — AVI BioPharma, Director, Clinical Operations
Locations (2):
- United Kingdom (2):
  - Great Ormond Street Hospital, London, England
  - Royal Victoria Infirmary, Newcastle upon Tyne, England

REFERENCES:
- [Result] Cirak S, Arechavala-Gomeza V, Guglieri M, Feng L, Torelli S, Anthony K, Abbs S, Garralda ME, Bourke J, Wells DJ, Dickson G, Wood MJ, Wilton SD, Straub V, Kole R, Shrewsbury SB, Sewry C, Morgan JE, Bushby K, Muntoni F. Exon skipping and dystrophin restoration in patients with Duchenne muscular dystrophy after systemic phosphorodiamidate morpholino oligomer treatment: an open-label, phase 2, dose-escalation study. Lancet. 2011 Aug 13;378(9791):595-605. doi: 10.1016/S0140-6736(11)60756-3. Epub 2011 Jul 23. PMID 21784508

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - 0.5 mg/kg/wk: Subjects in this group received a 0.5 mg/kg/wk dose of AVI-4658 over 12 weekly IV infusions in 50 mL of normal saline solution over a 60-minute period
Period: Overall Study
Arm/Group | Cohort 1 - 0.5 mg/kg/wk | Cohort 2 - 1.0 mg/kg/wk | Cohort 3 - 2.0 mg/kg/wk | Cohort 4 - 4.0 mg/kg/wk | Cohort 5 - 10.0 mg/kg/wk | Cohort 6 - 20.0 mg/kg/wk
Started | 4 | 2 | 2 | 3 | 4 | 4
Completed | 4 | 2 | 2 | 2 | 4 | 4
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 - 0.5mg/kg/wk: Subjects in this group received a 0.5 mg/kg/wk dose of AVI-4658 over 12 weekly IV infusions in 50 mL of normal saline solution over a 60-minute period
- Cohort 2 - 1.0mg/kg/wk: Subjects in this group received a 1.0 mg/kg/wk dose of AVI-4658 over 12 weekly IV infusions in 50 mL of normal saline solution over a 60-minute period
- Cohort 3 - 2.0mg/kg/wk: Subjects in this group received a 2.0 mg/kg/wk dose of AVI-4658 over 12 weekly IV infusions in 50 mL of normal saline solution over a 60-minute period
- Cohort 4 - 4.0mg/kg/wk: Subjects in this group received a 4.0 mg/kg/wk dose of AVI-4658 over 12 weekly IV infusions in 50 mL of normal saline solution over a 60-minute period
- Cohort 5 - 10.0mg/kg/wk: Subjects in this group received a 10.0 mg/kg/wk dose of AVI-4658 over 12 weekly IV infusions in 50 mL of normal saline solution over a 60-minute period
- Cohort 6 - 20.0mg/kg/wk: Subjects in this group received a 20.0 mg/kg/wk dose of AVI-4658 over 12 weekly IV infusions in 50 mL of normal saline solution over a 60-minute period
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - 0.5mg/kg/wk | Cohort 2 - 1.0mg/kg/wk | Cohort 3 - 2.0mg/kg/wk | Cohort 4 - 4.0mg/kg/wk | Cohort 5 - 10.0mg/kg/wk | Cohort 6 - 20.0mg/kg/wk | Total
Number analyzed (Participants) | 4 | 2 | 2 | 3 | 4 | 4 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.3 (0.50) | 6.0 (0.0) | 11.0 (2.83) | 9.7 (0.58) | 8.8 (2.75) | 8.8 (1.26) | 8.7 (1.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 4 | 2 | 2 | 3 | 4 | 4 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 2 | 2 | 3 | 4 | 4 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 1 | 2 | 3 | 4 | 4 | 18
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body Weight [Mean (Standard Deviation); unit: kilograms] | 33 (4.09) | 23.7 (3.46) | 42.6 (6.36) | 40.1 (19.00) | 34.6 (14.01) | 33.0 (8.71) | 34.5 (10.84)
Height [Mean (Standard Deviation); unit: centimeters] | 127.3 (5.05) | 110.7 (4.45) | 126.9 (5.09) | 126.9 (14.40) | 123.7 (10.04) | 126.5 (7.18) | 124.5 (8.99)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: Number of subjects with 1 or more Treatment Emergent Adverse Event that are possibly related to the investigational drug
Time Frame: Baseline to 6 months
Population: Safety Population - Any patient who received at least one dose of the study drug.
Measure: Number; unit: participants
Groups:
- Open Label Treatment Arm: AVI-4658 for Injection: AVI-4658 for Injection, is packaged as 100 mg/mL in phosphate buffered saline with 1 mL per vial. Study dosages will be infused over a 1 hour period with Normal saline as follows:
  Cohort 1: 0.5mg/kg once weekly for 12 weeks; Cohort 2: 1.0mg/kg once weekly for 12 weeks; Cohort 3: 2.0mg/kg once weekly for 12 weeks; Cohort 4: 4.0mg/kg once weekly for 12 weeks; Cohort 5: 10.0mg/kg once weekly for 12 weeks; Cohort 6: 20.0mg/kg once weekly for 12 weeks
Arm/Group | Open Label Treatment Arm
Number analyzed (Participants) | 19
participants | 14

2. Secondary Outcome: Pharmacokinetics - Mean Peak Plasma Concentration of AVI-4658 After Administration
Description: Standard Pharmacokinetic parameters estimated using non-compartmental modeling of plasma concentration data.
Time Frame: Samples were taken: 30 minutes pre dose; and at 5 (±1), 15 (±2), 30 (±5), 60 (±5), and 90 (±5) minutes; and 2, 4, 6, 8, 12, and 24 hours (all ± 15 minutes) post dose at Weeks 1, 6, and 12
Population: PK Evaluable Population: Included all patients who provided at least 1 PK sample. The reportable PK population included those patients with at least Cmax, Tmax, and AUC0-24 computed from 1 or more of the 3 sampling days (1st, 6th, 12th dose [Weeks 1, 6, and 12]).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Open Label Treatment Arm
Number analyzed (Participants) | 19
ng/mL | 39000 (16900)

3. Secondary Outcome: Efficacy of Eteplirsen Over 12 Weeks of Dosing
Description: Efficacy was defined as an estimated change in the percentage of dystrophin positive fibers (assessed by IHC) at Week 14 from Baseline after 12 weekly doses of eterplirsen. This outcome measure represents the number of patients to show an increase in the percentage of dystrophin-positive fibers.
Time Frame: Biopsies were taken at Baseline and Week 14
Population: Per Protocol Population - Included all patients who received all 12 doses of study treatment.
Measure: Number; unit: participants
Groups:
- Open Label Treatment Arm: Subjects will be sequentially allocated to one of 6 dose level cohorts and will receive 12 weekly IV infusions of AVI-4658 in 50 mL of normal saline solution over a 60-minute period
  AVI-4658 for Injection: AVI-4658 for Injection, is packaged as 100 mg/mL in phosphate buffered saline with 1 mL per vial. Study dosages will be infused over a 1 hour period with Normal saline as follows:
  Cohort 1: 0.5mg/kg once weekly for 12 weeks; Cohort 2: 1.0mg/kg once weekly for 12 weeks; Cohort 3: 2.0mg/kg once weekly for 12 weeks; Cohort 4: 4.0mg/kg once weekly for 12 weeks; Cohort 5: 10.0mg/kg once weekly for 12 weeks; Cohort 6: 20.0mg/kg once weekly for 12 weeks
Arm/Group | Open Label Treatment Arm
Number analyzed (Participants) | 17
participants | 11

4. Primary Outcome: Treatment Emergent Adverse Events
Description: Number of Patients with Treatment Emergent Adverse Events
Time Frame: from Baseline to Follow up (27 weeks)
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Open Label Treatment Arm
Number analyzed (Participants) | 19
participants | 19

5. Post Hoc Outcome: Adverse Events >15%
Description: Adverse events that occurred in >15% of overall patient population across dose level arms.
Time Frame: 27 Weeks
Population: Safety Population
Measure: Number; unit: Events
Groups:
- Cohort 1 - 0.5 mg/kg/wk: Subjects in this group received a 0.5 mg/kg/wk dose of AVI-4658 over 12 weekly IV infusions in 50 mL of normal saline solution over a 60 minute period
- Cohort 2 - 1.0 mg/kg/wk: Subjects in this group received a 1.0 mg/kg/wk dose of AVI-4658 over 12 weekly IV infusions in 50 mL of normal saline solution over a 60 minute period
- Cohort 3 - 2.0 mg/kg/wk: Subjects in this group received a 2.0 mg/kg/wk dose of AVI-4658 over 12 weekly IV infusions in 50 mL of normal saline solution over a 60 minute period
- Cohort 4 - 4.0 mg/kg/wk: Subjects in this group received a 4.0 mg/kg/wk dose of AVI-4658 over 12 weekly IV infusions in 50 mL of normal saline solution over a 60 minute period
- Cohort 5 - 10.0 mg/kg/wk: Subjects in this group received a 10.0 mg/kg/wk dose of AVI-4658 over 12 weekly IV infusions in 50 mL of normal saline solution over a 60 minute period
- Cohort 6 - 20.0 mg/kg/wk: Subjects in this group received a 20.0 mg/kg/wk dose of AVI-4658 over 12 weekly IV infusions in 50 mL of normal saline solution over a 60 minute period
Arm/Group | Cohort 1 - 0.5 mg/kg/wk | Cohort 2 - 1.0 mg/kg/wk | Cohort 3 - 2.0 mg/kg/wk | Cohort 4 - 4.0 mg/kg/wk | Cohort 5 - 10.0 mg/kg/wk | Cohort 6 - 20.0 mg/kg/wk
Number analyzed (Participants) | 4 | 2 | 2 | 3 | 4 | 4
Events
  Cardiomyopathy | 0 | 0 | 0 | 1 | 0 | 2
  Tachycardia | 0 | 0 | 0 | 1 | 0 | 2
  Abdominal Pain | 0 | 1 | 0 | 1 | 1 | 0
  Nausea | 0 | 0 | 1 | 1 | 0 | 1
  Vomiting | 0 | 0 | 1 | 1 | 1 | 0
  Influenza like illness | 0 | 0 | 2 | 0 | 1 | 0
  Rhinitis | 1 | 0 | 0 | 1 | 4 | 1
  Upper respiratory tract infection | 2 | 1 | 0 | 1 | 2 | 2
  Fall | 2 | 0 | 0 | 2 | 0 | 1
  Arthralgia | 1 | 0 | 1 | 1 | 0 | 0
  Back Pain | 1 | 0 | 1 | 2 | 2 | 1
  Myalgia | 1 | 1 | 1 | 0 | 1 | 0
  Dizziness | 0 | 0 | 1 | 1 | 0 | 1
  Headache | 2 | 1 | 2 | 0 | 2 | 1

ADVERSE EVENTS:
Time Frame: Adverse Event data for this study was collected from Baseline to Follow-up (27 Weeks)
Arm/Group | Cohort 1 - 0.5 mg/kg/wk | Cohort 2 - 1.0 mg/kg/wk | Cohort 3 - 2.0 mg/kg/wk | Cohort 4 - 4.0 mg/kg/wk | Cohort 5 - 10.0 mg/kg/wk | Cohort 6 - 20.0 mg/kg/wk
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2 | 1/2 | 1/3 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 2/2 | 2/2 | 3/3 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 0.5 mg/kg/wk (N=4) | Cohort 2 - 1.0 mg/kg/wk (N=2) | Cohort 3 - 2.0 mg/kg/wk (N=2) | Cohort 4 - 4.0 mg/kg/wk (N=3) | Cohort 5 - 10.0 mg/kg/wk (N=4) | Cohort 6 - 20.0 mg/kg/wk (N=4)
Post-Operative Nausea and Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture of Left Medial Malleolus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 0.5 mg/kg/wk (N=4) | Cohort 2 - 1.0 mg/kg/wk (N=2) | Cohort 3 - 2.0 mg/kg/wk (N=2) | Cohort 4 - 4.0 mg/kg/wk (N=3) | Cohort 5 - 10.0 mg/kg/wk (N=4) | Cohort 6 - 20.0 mg/kg/wk (N=4)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Platelet anisocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain - Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abasia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — One subject had a reduction in fractional shortening due DMD progression One subject had a deterioration of clinical signs of DMD
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incision site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heat Stroke (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetitie (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enuresis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the small number of study participants, a single adverse event (AE) in 1 patient exceeds the reporting threshold of 5%. Refer to the "Post-Hoc Outcome Measures" #5 for a summary of frequent and related AEs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI required written permission to publish any information relating to the trial and if given permission to acknowledge the sponsor's contribution and ownership of the materials.